CLINICAL TRIAL: NCT06790355
Title: Feasibility of Blood-based Test for Multi-cancer Early Detection in Asymptomatic Screening Population（ProSight）: a Multi-centre Interventional Study
Brief Title: ProSight: a Multi-centre Interventional Study Evaluating MCED in Asymptomatic Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Weihe Medical Laboratory Co., Ltd. (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Genie-ProSight
Record Dates: First submitted 2025-01-12; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer; Colorectal Cancer; Liver Cancer; Grastic Cancer; Esophageal Cancer
Keywords: multi-cancer early detection; MCED; cancer screening; circulating cell-free tumor DNA; methylation
MeSH Terms: conditions — Lung Neoplasms; Colorectal Neoplasms; Liver Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy subjects (Experimental)
  Interventions: Device: multi-cancer early detection

INTERVENTIONS:
Device: multi-cancer early detection — Blood collection for multi-cancer early detection（MCED）, followed by clinical diagnosis based on the results of MCED and standard-of-care screening

SUMMARY:
This is a prospective, multi-centre interventional study evaluating the feasibility of blood-based multi-cancer early detection test in asymptomatic screening cohort.

DETAILED DESCRIPTION:
Approximately 2527 participants will be enrolled and offered the multi-cancer early detection (MCED) test along with standard-of-care (SOC) cancer screenings and usual medical care. The investigational test is designed to detect five cancer types at a curable stage, which are lung cancer, colorectal cancer, liver cancer, gastric cancer and esophageal cancer. The test provides a binary result and predicts the signal origins if a cancer signal is detected. Those with "cancer signal detected" test results as well as those with warning signs of cancer during health check-up will undergo diagnostic procedures. The diagnostic work-up will be at the discretion of qualified oncologists, instead of being dictated by protocol.

Both the safety and performance of MCED in the screening setting will be evaluated. The extent of diagnostic testing, including laboratory and imaging tests and procedures required to achieve diagnostic resolution, will be recorded and assessed. Additionally, patient-reported outcomes relating to the testing experience will also be collected at specified time points using the Electronic Clinical Outcome Assessment (eCOA) app.

Participants will be actively followed for 1 year from the date of the blood draw.

ELIGIBILITY:
Inclusion Criteria:

* 40-74 years old
* Able to provide a written informed consent and willing to comply with all parts of the protocol procedures

Exclusion Criteria:

* With cancer-associated clinical symptoms or suspected of cancer within 30 days prior to screen
* Have definite contraindications of cancer screening examination and diagnostic procedures
* Unable to comply with the protocol procedures
* Personal history of cancer, diagnosed within the 3 years prior to expected enrollment date
* Have received or are undergoing curative cancer treatment within three years prior to recruitment. Adjuvant endocrinotherapy for cancer is not an exclusion criterion.
* Recipients of anti-tumor therapy within 30 days prior to screen
* Pregnancy or lactating women
* Recipients of organ transplant or prior bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 7 days prior to screen
* With autoimmune diseases
* Have an acute infection or inflammation or uncontrolled chronic infection within 14 days prior to blood draw
* Unsuitable for this trial determined by the researchers (eg. hemorrhagic diseases)

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2527 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of MCED in the intended use setting. | From enrollment to the Follow-up at 1 year
  Descriptive statistics will be used to summarize the number of 5 pre-specified cancers diagnosed by MCED.
Safety of MCED in the intended use setting. | From enrollment to the Follow-up at 1 year
  Descriptive statistics will be used to summarize the time to achieve diagnostic resolution following receipt of a positive MCED test and to assess the extent of testing pursued.

SECONDARY OUTCOMES:
Performance of MCED in the intended use setting. | From enrollment to the Follow-up at 1 year
  Positive Predictive Value defined as the proportion of participants with cancer diagnosis out of all participants with "signal detected" test result.
Cancer signal origin accuracy of MCED. | From enrollment to the Follow-up at 1 year
  Cancer signal origin accuracy defined as the proportion of participants with correct SCO predictions among those with positive test results who had a cancer diagnosis.
Clinical utility of MCED alongside SOC screening. | From enrollment to the Follow-up at 1 year
  Descriptive statistics will be used to summarize the number and types of cancers diagnosed by MCED among participants who are ineligible for SOC screening.
Participant-reported psychological impact. | From enrollment to the Follow-up at 1 year
  Changes in anxiety during study will be assessed using the short form of STAI (The state-trait anxiety inventory). Descriptive statistics for a total score will be used to measure feelings of anxiety.
Participant-reported health related quality of life (HRQoL) . | From enrollment to the Follow-up at 1 year
  Changes in HRQoL during study will be assessed using the EQ-5D-5L. Descriptive statistics for an index value at various time points will be used to reflect how good or bad a health state is.

OTHER OUTCOMES:
Participant-reported satisfaction with MCED. | From enrollment to the Follow-up at 1 year
  Descriptive statistics for a total score across all questions and individual ratings for each question.
Cross-reactivity of MCED. | From enrollment to the Follow-up at 1 year
  Descriptive statistics will be used to summarize the number and types of untrained cancers (beyond the 5 pre-specified cancers) diagnosed by MCED in participants for whom cancer signal origin directed workups do not result in diagnosis of cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, Principal Investigator — Fudan University; Xiaohui Wu, Study Director — Shanghai Weihe Medical Laboratory Co., Ltd.

IPD SHARING:
Plan to Share IPD: No